CLINICAL TRIAL: NCT01597700
Title: A RANDOMIZED, BALANCED, OPEN LABEL, CROSSOVER, TWO PERIOD, TWO TREATMENT, TWO SEQUENCE, SINGLE DOSE, BIOEQUIVALENCE STUDY OF ACOTRAL® EZETIMIBE 10 MG TABLETS CONTAINING EZETIMIBE MANUFACTURED BY LABORATORIOS PHOENIX S.A.I.C.F, ARGENTINA AND ZETIA® EZETIMIBE 10 MG TABLETS OF MERCK/SCHERING - PLOUGH PHARMACEUTICALS, USA IN HEALTHY ADULT HUMAN MALE SUBJECTS UNDER FASTING CONDITION
Brief Title: Acotral® Versus Zetia® Ezetimibe Bioequivalance Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116051
Record Dates: First submitted 2012-03-22; First posted 2012-05-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acotral® ezetimibe 10mg (Experimental): Subjects will be fasted overnight and receive one tablet by mouth in accordance with a randomisation list and venous blood samples will be taken at specified intervals over the ensuing 3 day.
  Interventions: Drug: 10mg Ezetimibe
- Zetia® ezetimibe 10mg (Active Comparator): Subjects will be fasted overnight and receive one tablet by mouth in accordance with a randomisation list and venous blood samples will be taken at specified intervals over the ensuing 3 days.
  Interventions: Drug: 10 mg Ezetimibe - wash out period

INTERVENTIONS:
Drug: 10mg Ezetimibe — 1 tablet taken by mouth
  Arms: Acotral® ezetimibe 10mg
Drug: 10 mg Ezetimibe - wash out period — 1 tablet taken by mouth received after wash out period
  Arms: Zetia® ezetimibe 10mg

SUMMARY:
Bioequivalence study comparing test Acotral® ezetimibe 10 mg tablet manufactured by Laboratorios Phoenix, with a reference comparator Zetia® ezetimibe 10 mg tablet of Merck/Schering-Plough Pharmaceuticals. The CRO Clinigene Bangalore, will conduct the study. Fifty two healthy adult subjects who have satisfied the inclusion and exclusion criteria and given their informed consent will be entered into the study. They will be fasted and receive one tablet by mouth in accordance with a randomisation list and blood samples will be taken at specified intervals over the ensuing 3 days. Between 14 and 21 days later, subjects will receive the opposite tablet and the clinical process repeated. Subjects will be continuously monitored while in the trial clinic and at ambulatory visits with regular measurements of vital signs and questioned for adverse events. Drug concentrations will be analysed and these results compared to ascertain bioequivalence by applying statistical methods to the pharmacokinetic data; this information and all safety data will be formally reported.

DETAILED DESCRIPTION:
This is a randomized, balanced, open label, crossover, two period, two treatment, two sequence, single dose bioequivalence study comparing test Acotral® ezetimibe 10 mg tablet manufactured by Laboratorios Phoenix, Argentina with a reference comparator Zetia® ezetimibe 10 mg tablet of Merck/Schering-Plough Pharmaceuticals, USA. The CRO Clinigene International Ltd, Bangalore, India will conduct the study. Fifty two healthy male adult subjects who have satisfied the inclusion and exclusion criteria and given their written informed consent will be entered into the study. They will be fasted overnight and receive one tablet by mouth in accordance with a randomisation list and venous blood samples will be taken at specified intervals over the ensuing 3 days; meals and water ad libitum will be allowed. Between 14 and 21 days later, subjects will return to the clinic and follow the same procedure to receive the opposite tablet and the clinical process repeated. Subjects will be continuously safety monitored while in the trial clinic and at ambulatory visits with regular measurements of vital signs and questioned for adverse events in accordance with the trial clinic SOPs. Drug concentrations will be analysed and these results compared in accordance with the study protocol to ascertain bioequivalence by applying statistical methods to the pharmacokinetic data; this information and all safety data will be formally reported to GSK.

ELIGIBILITY:
Inclusion Criteria:

* Literate healthy adult male human subjects within the age range of 18 to 45 years inclusive.
* Weight not less than 50 kg.
* Normal BMI [18.5 to 24.99 kg/m2 inclusive].
* Willingness to provide written informed consent to participate in the study and capable of giving written informed consent to participate in the study.
* Free of significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12-lead ECG, Chest X-ray [PA view].
* AST, ALT, alkaline phosphatase and bilirubin 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Absence of disease markers of HIV 1 and 2, Hepatitis B and C and Syphilis.
* ECG normal for morphology and measurements. QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* History or presence of significant: Cardiovascular, pulmonary, hepatic, renal, hematological, gastro-intestinal, endocrine, immunologic, dermatologic, neurological, psychiatric disease.
* History or presence of significant:
* Alcohol dependence, alcohol abuse during past one year.
* Drug abuse for the last one month and other illicit drugs for the last 6 months.
* Smoking of more than 5 cigarettes per day or consumption of other forms of tobacco containing products.
* Asthma, urticaria or other allergic type reactions after taking aspirin or any other drug.
* Ulceration or history of gastric and / or duodenal ulcer.
* Jaundice in the past 6 months.
* Bleeding disorder.
* Allergy to the test drug or any drug chemically similar to the drug or to the excipients of the products under investigation.
* Donation of 500 mL blood within 08 weeks prior to receiving the first dose of study drug.
* Subjects who have participated in another clinical study in the past 3 months prior to commencement of this study.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study assessments or compromise subject safety.
* Any difficulty in accessibility of forearm veins for cannulation or blood sampling.
* Refuse to abstain from food for at least 10 h prior to drug administration and for at least 4 h after dose in each period.
* Refuse to abstain from fluid for at least 1 h prior to and until 1 h post each dose.
* Found positive in breath alcohol test done on the day of check-in and ambulatory visit.
* Found positive in urine test for drug of abuse done on the day of check-in.
* History of difficulty in swallowing tablet.
* Use of enzyme modifying drugs within 30 days prior to receiving the first dose of study medication.
* Other Eligibility Criteria Considerations
* To assess any potential impact on subject eligibility with regard to safety, the investigator must refer to the product data sheet for detailed information regarding warnings, precautions, contraindications, adverse events, and other significant data pertaining to the product being used in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01-13 (Actual); Primary Completion 2012-01-30 (Actual); Study Completion 2012-01-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in plasma ezetimibe concentrations in time after dosing | At 0 time and up to 72 hours after last dose
  Liquid chromatography and mass spectrometry
Number of participants with adverse events | At 0 time and up to 72 hours after last dose
  Safety monitoring
Number of participants with changes in haematology and/or chemistry | 21 to 0 days before first dose and 3 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Electronics City, Bengalore, India

REFERENCES:
- See also: Results for study 116051 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116051?search=study&search_terms=116051#rs